CLINICAL TRIAL: NCT03744234
Title: Platelet-rich Plasma in the Sacroiliac Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAQ8843
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Sacroiliac Joint Arthritis
Keywords: PRP; Platelet-Rich Plasma; Sacroiliac Joint Pain; SIJ Pain; Osteoarthritis
MeSH Terms: conditions — Sacroiliitis; Osteoarthritis | interventions — Steroids

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-Rich Plasma Injection (Experimental): Autologous injection of platelet-rich plasma (PRP) in the sacroiliac joint
  Interventions: Procedure: PRP
- Steroid Injection (Active Comparator): Steroid injection in the sacroiliac joint
  Interventions: Procedure: Steroid Injection

INTERVENTIONS:
Procedure: PRP — Autologous platelet-rich plasma
  Arms: Platelet-Rich Plasma Injection
Procedure: Steroid Injection — Steroid injection
  Arms: Steroid Injection

SUMMARY:
This is a double-blinded study where the injecting physicians and the patients will not know which arm they are randomized to. Each participant will be followed up for 6 months following the injection, and will have in office visits at the injection and approximately 2 weeks post injection. They will be called at month 1, 3, and 6 post injection to assess for any adverse events and number of physical therapy hours or changes in medication. At time of injection, 2 weeks post, and 1, 3 and 6 months after they will be asked to answer some questionnaires on pain and function.

DETAILED DESCRIPTION:
Sacroiliac joint (SIJ) pain is a common and significant source of chronic low back pain. It has been broadly defined as pain located in the area of the SIJ that can be elicited by various pain provocation tests and relieved after infiltration of the joint with local anesthetic.

Essentially, a patients own blood is collected and spun at varying speeds until it separates into 3 layers, one of which is the platelet-rich plasma. Platelet-rich plasma (PRP) injections are commonly used in various conditions including chronic tendinopathy, soft tissue injuries, and ligamentous injuries. More recently, there has been a greater interest in examining the efficacy of PRP as a treatment for musculoskeletal conditions affecting joints, such as osteoarthritis (OA). To the investigators' knowledge, there are currently no reported studies evaluating the efficacy of PRP for SIJ pain. Given the previously discussed application and evidence behind the use of PRP in the knee and hip joints, the investigators propose that PRP can also provide a similar solution for treating SIJ pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Sacroiliac/Lower back pain
* Positive block
* Eligible for steroid injection
* Positive physical manual assessments

Exclusion Criteria:

* Steroid allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Pain (VAS) Score | Up to 6 months
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Change in Score on the Oswestry Low Back Pain Disability Questionnaire | Up to 6 months
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) allows researchers and disability evaluators to measure a patient's permanent functional disability. For each section the total possible score is 5 (0= no pain to 5=worst pain) and there are 10 sections of questions. An aggregate score (percentage) is then calculated, with 0% indicating no disability to 100%, indicating crippled or bed-bound.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. Solberg, DO, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen AS, Solberg J, Smith C, Chi M, Lowder R, Christolias G, Singh JR. Intra-Articular Platelet Rich Plasma vs Corticosteroid Injections for Sacroiliac Joint Pain: A Double-Blinded, Randomized Clinical Trial. Pain Med. 2022 Jul 1;23(7):1266-1271. doi: 10.1093/pm/pnab332. PMID 34850180